CLINICAL TRIAL: NCT06404398
Title: Clinical Evaluation of Single Versus Multi-Shade Direct Composite Resin Veneers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Abd El Ghany Mohammed, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Direct Composite Resin Veneers
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-05

CONDITIONS: Tooth Discoloration
Keywords: OMNICHROMA; Veneers; USPHS criteria
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical study
Who Masked: Participant, Outcomes Assessor
Masking Description: This clinical study was double-blind study as the evaluators who were not included in the restorative procedures and the patients were blinded to tested groups, but the operator wasn't blinded to these groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMNICHROMA (Experimental): one single shade
  Interventions: Other: OMNICHROMA, Ceram. x spectra
- Ceram. x spectra (Experimental): multi- shade
  Interventions: Other: OMNICHROMA, Ceram. x spectra

INTERVENTIONS:
Other: OMNICHROMA, Ceram. x spectra — Each patient had two types of veneers.

SUMMARY:
The aim of this study was to clinically evaluate single and multi-shade direct veneers.

DETAILED DESCRIPTION:
The use of direct, light-activated resin composites in esthetic restorative dentistry has grown dramatically in response to growing needs. Recent developments have resulted in the creation of restorative materials and methods that, particularly in the anterior area, attempt to restore the natural appearance of the teeth.

Numerous clinical conditions, including tooth discolorations, severe fractures, misaligned teeth, and dental caries lesions, can significantly affect smile harmony and esthetic appearance, which can lower quality of life.

Modern cosmetic dentistry began with the introduction of laminate veneers in the 1970s, which combined the ideas of tooth conservation and aesthetics. Because laminate veneers (LVs) offer the potential to satisfy the need for extremely beautiful, minimally invasive, long-lasting restorations with superior clinical performance, they have gained popularity as a treatment option.

Direct composite veneering preserves natural tooth structure, may be completed chairside, doesn't require repeated appointments, doesn't require luting agents, is minimally invasive, readily repaired, and is less expensive because there are no laboratory fees. Furthermore, their abrasion rates are comparable to those of real tooth structures.

ELIGIBILITY:
Inclusion Criteria:

* Good hygiene.
* Vital discolored anterior teeth

Exclusion Criteria:

* severe discoloration
* Para functional activities
* Non-vital teeth.
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
assess single and multi-shade direct composite resin veneers | 18 months evaluation periods
  Two evaluators assessed the restorations based on modified United States Public Health Service criteria. Score(0) represents ideal clinical scenario, Score(1) acceptable, Score (2) satisfactory, and Score(3) and Score (4) considered clinically unsatisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- Restorative Department, Faculty of Dentistry, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blatz MB, Chiche G, Bahat O, Roblee R, Coachman C, Heymann HO. Evolution of Aesthetic Dentistry. J Dent Res. 2019 Nov;98(12):1294-1304. doi: 10.1177/0022034519875450. PMID 31633462
- [Result] Araujo E, Perdigao J. Anterior Veneer Restorations - An Evidence-based Minimal-Intervention Perspective. J Adhes Dent. 2021 Apr 7;23(2):91-110. doi: 10.3290/j.jad.b1079529. PMID 33825424
- [Result] Akgul S, Gundogdu C, Bala O. Effects of storage time and restoration depth on instrumental color adjustment potential of universal resin composites. J Oral Sci. 2022 Jan 19;64(1):49-52. doi: 10.2334/josnusd.21-0290. Epub 2021 Dec 15. PMID 34911896
- [Result] Chen F, Toida Y, Islam R, Alam A, Chowdhury AFMA, Yamauti M, Sano H. Evaluation of shade matching of a novel supra-nano filled esthetic resin composite employing structural color using simplified simulated clinical cavities. J Esthet Restor Dent. 2021 Sep;33(6):874-883. doi: 10.1111/jerd.12671. Epub 2020 Nov 14. PMID 33188588
- [Result] Attia YS, Sherif RM, Zaghloul HH. Survival of Hybrid Laminate Veneers using two different tooth preparation techniques: Randomized Clinical Trial. Braz Dent J. 2021 Nov-Dec;32(6):36-53. doi: 10.1590/0103-6440202103907. PMID 35019018
- [Result] Fahl N Jr,, Ritter AV. Composite veneers: The direct-indirect technique revisited. J Esthet Restor Dent. 2021 Jan;33(1):7-19. doi: 10.1111/jerd.12696. Epub 2020 Dec 18. PMID 33336852
- [Result] Gresnigt MMM, Cune MS, Jansen K, van der Made SAM, Ozcan M. Randomized clinical trial on indirect resin composite and ceramic laminate veneers: Up to 10-year findings. J Dent. 2019 Jul;86:102-109. doi: 10.1016/j.jdent.2019.06.001. Epub 2019 Jun 7. PMID 31181242
- [Result] Kam Hepdeniz O, Temel UB. Clinical survival of No-prep indirect composite laminate veneers: a 7-year prospective case series study. BMC Oral Health. 2023 May 3;23(1):257. doi: 10.1186/s12903-023-02949-5. PMID 37138297
- [Result] Haak R, Bruckner A, Hafer M, Scholz M, Schneider H. Is There an Association Between Clinical and SEM Quantitative Marginal Analysis in a 90-month Trial? J Adhes Dent. 2021;23(1):37-46. doi: 10.3290/j.jad.b916821. PMID 33512114
- [Result] Ojeda G D, Naves LZ, Oosterhaven A, Kleinsman R, Baumer-Konig A, Korner G, Wendler M, Gresnigt M. 8-year multicenter retrospective study on partial laminate veneers. J Prosthodont Res. 2023 Apr 12;67(2):206-213. doi: 10.2186/jpr.JPR_D_22_00079. Epub 2022 Jul 5. PMID 35793984
- [Result] Ahmed MA, Jouhar R, Khurshid Z. Smart Monochromatic Composite: A Literature Review. Int J Dent. 2022 Nov 8;2022:2445394. doi: 10.1155/2022/2445394. eCollection 2022. PMID 36398065
- [Result] Yagci O, Fidan M. Influence of Thickness on the Translucency Parameter and Whiteness Index of Single-Shade Resin Composites. Oper Dent. 2024 Mar 1;49(2):189-199. doi: 10.2341/23-053-L. PMID 38349843
- [Result] Korkut B, Unal T, Can E. Two-year retrospective evaluation of monoshade universal composites in direct veneer and diastema closure restorations. J Esthet Restor Dent. 2023 Apr;35(3):525-537. doi: 10.1111/jerd.12992. Epub 2022 Dec 7. PMID 36478098
- [Result] Hayashi S, Homma S, Takanashi T, Hirano T, Yoshinari M, Yajima Y. Wear properties of esthetic dental materials against translucent zirconia. Dent Mater J. 2019 Mar 31;38(2):250-256. doi: 10.4012/dmj.2018-133. Epub 2018 Dec 11. PMID 30541995
- [Result] Yilmaz Atali P, Dogu Kaya B, Manav Ozen A, Tarcin B, Senol AA, Tuter Bayraktar E, Korkut B, Bilgin Gocmen G, Tagtekin D, Turkmen C. Assessment of Micro-Hardness, Degree of Conversion, and Flexural Strength for Single-Shade Universal Resin Composites. Polymers (Basel). 2022 Nov 17;14(22):4987. doi: 10.3390/polym14224987. PMID 36433113
- [Result] Hampe-Kautz V, Salehi A, Senger B, Etienne O. A comparative in vivo study of new shade matching procedures. Int J Comput Dent. 2020;23(4):317-323. PMID 33491927